CLINICAL TRIAL: NCT04329169
Title: Digital Assessment of a Full Digital Implant-Prosthetic Workflow for a Prefabricated Single Implant-Supported Restoration (A Clinical Trial)
Brief Title: Digital Assessment of a Full Digital Implant-Prosthetic Workflow for a Prefabricated Single Implant-Supported Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Dental Public Health clinical instructor and study statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Virtual implant planning
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Implant Planning (Experimental)
  Interventions: Other: Virtual Implant Planning

INTERVENTIONS:
Other: Virtual Implant Planning — According to the virtual implant plan, a CAD/CAM tooth supported surgical guide will be fabricated to place the dental implant with a fully guided surgical protocol.The surgical guide will be manufactured from a photopolymer resin using a 3D printing machine. A hex- shaped metal sleeve will be inserted in the surgical guide with the flat surface located buccally so that it will help in orientation of the implant hex during the implant placement.

SUMMARY:
The aim of the present study was to evaluate the accuracy of a prefabricated digitally planned provisional restoration on a single- implant placed with a fully guided surgical protocol.

DETAILED DESCRIPTION:
Fifteen dental implants were placed in partially edentulous patients with single bounded lower posterior edentulous area selected from those admitted to the Prosthodontics Department, Faculty of Dentistry, Alexandria University. A full digital implant-prosthetic protocol was followed and a quantitative evaluation of the accuracy of the protocol was performed using computer software and superimposition of the planned and post-operative images was done.

ELIGIBILITY:
Inclusion Criteria:

* Patients missing lower first molar unilaterally or bilaterally.
* Presence of full or nearly full complement of opposing natural teeth.

Exclusion Criteria:

* If teeth adjacent to the planned implant site showed infections, endodontic or periodontal problems.
* Patients with a debilitating systemic disease, bone diseases, radiotherapy or chemotherapy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
3D- Deviation of the implant | 3 months
  The 3D deviation will be calculated by a software taking into consideration the deviation on each direction set as follows: x= buccolingual error, y= mesiodistal error, and z= apicocoronal error, using Pythagorean Theorem: 3D deviation= square root of (x squared + y squared + z squared)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Badee, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mariam Bahgat, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Haitham Ismail, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Yassmin Tahamawy, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Naema Ammar, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt